CLINICAL TRIAL: NCT02146027
Title: Immunological Effects of Continuous, Once a Day Use of Lactobacillus Casei Shirota on HIV-infected Patients on Suppressive Antiretroviral Treatment With Poor CD4+ T-cell Recovery
Brief Title: Once a Day Use of Lactobacillus Casei Shirota on HIV-infected Patients Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Principal Investigator, Esper Georges Kallás, MD PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: YAKULT
Record Dates: First submitted 2014-02-18; First posted 2014-05-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; Lactobacillus casei Shirota; NK cell; CD4; Lymphocyte; Cell activation; Antiretroviral therapy; Immune discordants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fermented Milk Drink Yakult 40 (Experimental): Lactobacillus casei Shirota, contained in the Fermented Milk Drink Yakult 40
  Once daily Lactobacillus casei Shirota, with 40 billion bacteria per 80 g (concentration of 5 x 10^8 CFU/g). Intervention will be used for 12 weeks.
  Interventions: Dietary Supplement: Fermented Milk Drink Yakult 40
- Placebo (Placebo Comparator): The placebo would be an analogous product without Live Lactic Bacteria (Lactobacillus casei Shirota) presented in the same bottle and similar flavor.
  Both, Yakult 40 and placebo should be stored refrigerated between 1° and 10°C and
  Interventions: Dietary Supplement: Fermented Milk Drink Yakult 40

INTERVENTIONS:
Dietary Supplement: Fermented Milk Drink Yakult 40 — Lactobacillus casei Shirota, with 40 billion bacteria per 80 g (concentration of 5 x 10^8 CFU/g). Intervention will be used for 12 weeks.
  Other Names: Yakult; Live Lactic Bacteria (Lactobacillus casei Shirota)
Dietary Supplement: Fermented Milk Drink Yakult 40 — Ingredients: Skimmed milk and/or Reconstituted Skimmed Milk, Sugar, Glucose, Live Lactic Bacteria (Lactobacillus casei Shirota) 40 billions per 80 g - concentration of 5 x 108 CFU/g), Flavour. Gluten Free.
  Other Names: Live Lactic Bacteria (Lactobacillus casei Shirota); Yakult

SUMMARY:
In this study, HIV-infected patients with poor recovery of CD4+ T cells and successful viral control after treatment with antiretroviral therapy will be enrolled to receive once a day Lactobcillus casei Shirota or placebo in a double-blind, randomized fashion. Immune parameters will be monitored for 12 weeks in both arms.

The main outcome is CD4+ T cell recovery. Secondary outcomes will include NK cells and T cells immune parameters.

DETAILED DESCRIPTION:
In this study, HIV-infected patients with poor recovery of CD4+ T cells and successful viral control after treatment with antiretroviral therapy will be enrolled to receive once a day Lactobcillus casei Shirota or placebo in a double-blind, randomized fashion.

The main objective is to investigate whether the continuous, once a day, 12-weeks use of Yakult product containing Lactobacillus casei Shirota could affect immunological parameters in HIV-infected patients on suppressive antiretroviral treatment with poor CD4+ T cell recovery. A total of 48 volunteers will be followed for 12 week after initiation of daily use of Lactobcillus casei Shirota or placebo, randomized in a 1:1 ratio.

We hypothesize that use of the Yakult product containing Lactobacillus casei Shirota after 12 weeks of continuous use will increase the level of CD4+ T-cells, at least, 50 cells/mm³.

We also propose to investigate several markers of immune response, including T cellular activation and NK cells function, and changes in the intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Male or female HIV-1 infected patients aged between 18 and 60 years.
* Patient on suppressive antiretroviral treatment with poor CD4+ T-cell recovery.
* No change in antiretroviral therapy in the last six months or intended change in the next 12 weeks.
* Availability for the study procedures during the study period.
* Giving informed consent to participate in the study

Exclusion Criteria:

* Diagnosis of any concomitant infections or diseases that might affect immunity or natural history of HIV-1 infection including active Hepatitis B infection, Hepatitis C infection, diabetes mellitus, neoplasias and autoimmune diseases.
* Use of treatments that might affect immunity in the last four weeks including immunomodulators, corticosteroids (only systemic use for two weeks or more), or antineoplasic agents.
* History of intolerance or allergy to cow milk or any other component of the study product including lactose intolerance, casein allergy, etc.
* Pregnancy, nursing mother or intention of became pregnant during the study period (only female participants).
* Unable to safely store the study product at home in the conditions recommended by the manufacturer.
* Any other condition that might interfere with the study procedure according to the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Increase between baseline and after 6 weeks and 12 weeks in the absolute CD4+ T-cell count in active and placebo group. | 12 weeks
  Only differences greater than 50 T CD4+ cells/mm³ would be included in the analysis.

SECONDARY OUTCOMES:
Change from baseline in level of cell activation at week 12 count | baseline, week 12
  Cell activation will be accessed by flow cytometry assays in a FACSCanto flow cytometer, using the following monoclonal antibodies: CD3, CD4, CD8, CD38, CCR5, CD69, anti-HLA-DR+
Change from baseline in level of cell activation at week 6 | baseline, week 6
  Cell activation will be accessed by flow cytometry assays in a FACSCanto flow cytometer, using the following monoclonal antibodies: CD3, CD4, CD8, CD38, CCR5, CD69, anti-HLA-DR+
Change from baseline in NK cytototoxic activity against K562 cells at week 6 | baseline, week 6
  NK cell phenotyping and function will be assessed according to Long et al., were subpopulations of NK cells will be assessed by the expression of CD56, CD16 molecules in the CD3-CD14-CD20- population of mononuclear cells. Production of IFNgama and CD103a proteins will be evaluated by flow cytometry in K562 stimulated mononuclear cells
Change from baseline in NK cytototoxic activity against K562 cells at week 12 | baseline, week 12
  NK cell phenotyping and function will be assessed according to Long et al., were subpopulations of NK cells will be assessed by the expression of CD56, CD16 molecules in the CD3-CD14-CD20- population of mononuclear cells. Production of IFNgama and CD103a proteins will be evaluated by flow cytometry in K562 stimulated mononuclear cells
Change from baseline in Intestinal symptoms score of the Inflammatory Bowel Disease Questionnaire (IBQD) at week 12 | baseline, week 12
Change from baseline in the intestinal microbiome in the participants taking Lactobacillus casei Shirota at week 12 | baseline, week 12
Number of participants with adverse events reasonable causal relationship with the study product in active and placebo groups | 12 weeks
Change from baseline in plasma sCD4 levels at week 6 | baseline, week 6
  CD14 levels will be measured using commercially available kits
Change from baseline in plasma sCD4 levels at week 12 | baseline, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Esper G Kallás, MD PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo - General Hospital, São Paulo, Brazil

REFERENCES:
- [Result] Boyle RJ, Robins-Browne RM, Tang ML. Probiotic use in clinical practice: what are the risks? Am J Clin Nutr. 2006 Jun;83(6):1256-64; quiz 1446-7. doi: 10.1093/ajcn/83.6.1256. PMID 16762934
- [Result] Brenchley JM, Douek DC. HIV infection and the gastrointestinal immune system. Mucosal Immunol. 2008 Jan;1(1):23-30. doi: 10.1038/mi.2007.1. PMID 19079157
- [Result] Corazza GR, Ginaldi L, Furia N, Marani-Toro G, Di Giammartino D, Quaglino D. The impact of HIV infection on lactose absorptive capacity. J Infect. 1997 Jul;35(1):31-5. doi: 10.1016/s0163-4453(97)90905-1. PMID 9279721
- [Result] Fujimori S, Gudis K, Mitsui K, Seo T, Yonezawa M, Tanaka S, Tatsuguchi A, Sakamoto C. A randomized controlled trial on the efficacy of synbiotic versus probiotic or prebiotic treatment to improve the quality of life in patients with ulcerative colitis. Nutrition. 2009 May;25(5):520-5. doi: 10.1016/j.nut.2008.11.017. Epub 2009 Feb 8. PMID 19201576
- [Result] Hummelen R, Vos AP, van't Land B, van Norren K, Reid G. Altered host-microbe interaction in HIV: a target for intervention with pro- and prebiotics. Int Rev Immunol. 2010 Oct;29(5):485-513. doi: 10.3109/08830185.2010.505310. PMID 20839912
- [Result] Irvine SL, Hummelen R, Hekmat S, Looman CW, Habbema JD, Reid G. Probiotic yogurt consumption is associated with an increase of CD4 count among people living with HIV/AIDS. J Clin Gastroenterol. 2010 Oct;44(9):e201-5. doi: 10.1097/MCG.0b013e3181d8fba8. PMID 20463586
- [Result] Marchetti G, Bellistri GM, Borghi E, Tincati C, Ferramosca S, La Francesca M, Morace G, Gori A, Monforte AD. Microbial translocation is associated with sustained failure in CD4+ T-cell reconstitution in HIV-infected patients on long-term highly active antiretroviral therapy. AIDS. 2008 Oct 1;22(15):2035-8. doi: 10.1097/QAD.0b013e3283112d29. PMID 18784466
- [Result] Marchetti G, Cozzi-Lepri A, Merlini E, Bellistri GM, Castagna A, Galli M, Verucchi G, Antinori A, Costantini A, Giacometti A, di Caro A, D'arminio Monforte A; ICONA Foundation Study Group. Microbial translocation predicts disease progression of HIV-infected antiretroviral-naive patients with high CD4+ cell count. AIDS. 2011 Jul 17;25(11):1385-94. doi: 10.1097/QAD.0b013e3283471d10. PMID 21505312
- [Result] Massanella M, Negredo E, Perez-Alvarez N, Puig J, Ruiz-Hernandez R, Bofill M, Clotet B, Blanco J. CD4 T-cell hyperactivation and susceptibility to cell death determine poor CD4 T-cell recovery during suppressive HAART. AIDS. 2010 Apr 24;24(7):959-68. doi: 10.1097/QAD.0b013e328337b957. PMID 20177358
- [Result] Piketty C, Castiel P, Belec L, Batisse D, Si Mohamed A, Gilquin J, Gonzalez-Canali G, Jayle D, Karmochkine M, Weiss L, Aboulker JP, Kazatchkine MD. Discrepant responses to triple combination antiretroviral therapy in advanced HIV disease. AIDS. 1998 May 7;12(7):745-50. doi: 10.1097/00002030-199807000-00011. PMID 9619806
- [Result] Rajasuriar R, Booth D, Solomon A, Chua K, Spelman T, Gouillou M, Schlub TE, Davenport M, Crowe S, Elliott J, Hoy J, Fairley C, Stewart G, Cameron P, Lewin SR. Biological determinants of immune reconstitution in HIV-infected patients receiving antiretroviral therapy: the role of interleukin 7 and interleukin 7 receptor alpha and microbial translocation. J Infect Dis. 2010 Oct 15;202(8):1254-64. doi: 10.1086/656369. PMID 20812848
- [Result] Trois L, Cardoso EM, Miura E. Use of probiotics in HIV-infected children: a randomized double-blind controlled study. J Trop Pediatr. 2008 Feb;54(1):19-24. doi: 10.1093/tropej/fmm066. Epub 2007 Sep 17. PMID 17878180
- [Result] Tinmouth J, Kandel G, Tomlinson G, Walmsley S, Steinhart AH, Glazier R. The effect of dairy product ingestion on human immunodeficiency virus-related diarrhea in a sample of predominantly gay men: a randomized, controlled, double-blind, crossover trial. Arch Intern Med. 2006 Jun 12;166(11):1178-83. doi: 10.1001/archinte.166.11.1178. PMID 16772244
- [Result] Woelk CH, Beliakova-Bethell N, Goicoechea M, Zhao Y, Du P, Rought SE, Lozach J, Perez-Santiago J, Richman DD, Smith DM, Little SJ. Gene expression before HAART initiation predicts HIV-infected individuals at risk of poor CD4+ T-cell recovery. AIDS. 2010 Jan 16;24(2):217-22. doi: 10.1097/QAD.0b013e328334f1f0. PMID 19952713